CLINICAL TRIAL: NCT02851550
Title: Assessement of the Prevalence of Lysosomal Acid Lipase Deficiency in Liver Post-transplant Patients
Acronym: LALTH-2
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Hospices Civils de Lyon (Other)
Responsible Party: Sponsor
Other Study IDs: 69HCL16_0485
Record Dates: First submitted 2016-07-28; First posted 2016-08-01 (Estimated); Last update posted 2016-08-01 (Estimated); Status verified 2016-07

CONDITIONS: Liver Post-transplant Patients
Keywords: liver; transplant; Lysosomal Acid Lipase
MeSH Terms: conditions — Cholesterol Ester Storage Disease

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — Few drops of blood absorbed onto blotting paper for enzymatic analysis

SUMMARY:
Lysosomal Acid Lipase (LAL) deficiency is a rare, autosomal recessive storage disease linked to decrease enzymatic activity of LAL, responsible for intracellular accumulation of cholesterol esters and triglycerides.

The accumulation of lipid is in hepatocytes, Kupffer cells and macrophages leading to a fatty liver, hepatic fibrosis that can evolve up to cirrhosis.

LAL deficiency is responsible for significant morbidity and early mortality in children, adolescents and adults in connection with a multi visceral disease reaching the liver, gastrointestinal tract and the vascular endothelium. The disease is caused by homozygous or heterozygous mutations in the gene (LIPA chromosome 10q23.2-23.3) which is responsible for the synthesis of the LAL.

The disease can be diagnosed by enzymatic analysis using few drops of blood absorbed onto blotting paper.

Patients with this deficiency LAL, have no or reduced activity of this enzyme. Because of its rarity, the deficit in LAL is under diagnosed or is diagnosed in patients with liver biological disturbances and / or lipid profile disturbances, steatohepatitis-hepatitis (NASH), the steatosis (NAFLD), the cryptogenic cirrhosis or Wilson disease.

Inclusion period of 12 to 18 months (100 patients).

ELIGIBILITY:
Inclusion Criteria:

* liver post-transplant patient
* patients with cryptogenic cirrhosis, NASH

Exclusion Criteria:

* Patients without metabolic syndrome clinical, biological or radiological.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The Assessment of the prevalence of Lysosomal Acid Lipase deficiency were performed from few blood drops absorbed onto blotting paper during a routine visit in liver post-transplant patients Patients will be included after liver transplantation. The enzymatic analysis onto blotting paper will be made during a routine visit in patients with cryptogenic cirrhosis, NASH (isolated or associated with other liver disease).
  Oral and written information will be given by the clinician. Only research team members will have access to patient data and their analysis. The patient data (age, gender, medical history, etiology of liver disease, liver function, lipid, glucose, radiological ...) will be collected and stored in an Excel file.
  The diagnosis analysis deficit LAL will be performed as described in the article by Hamilton.
Sampling Method: Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2015-12; Primary Completion 2017-12 (Estimated); Study Completion 2018-06 (Estimated)

PRIMARY OUTCOMES:
Prevalence of Lysosomal Acid Lipase deficiency in liver post-transplant patients | During the routine visit (Day 1)
  Assessment of the prevalence of Lysosomal Acid Lipase deficiency in liver post-transplant patients

CONTACTS AND LOCATIONS:
Overall Officials: Sylvie Radenne, MD, Principal Investigator — Hospices Civils de Lyon
Locations (1):
- Hépato-Gastro-Entérologie, Hôpital de la Croix Rousse, 103 gde rue de la Croix Rousse, Lyon, France